CLINICAL TRIAL: NCT04143607
Title: A Phase III,Double-Blind, Randomised Study to Assess the Efficacy and Safety of ASK120067 Versus Gefitinib as First-Line Treatment in Patients With Epidermal Growth Factor Receptor Mutation Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: ASK120067 Versus Gefitinib as First-line Treatment for EGFRm Locally Advanced or Metastatic NSCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASK-LC-120067-F-III
Record Dates: First submitted 2019-10-12; First posted 2019-10-29 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Intervention Model Description: Triple (Participant, Investigator, Outcomes Assessor)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASK120067+ placebo Gefitinib (Experimental): ASK120067 (80 mg orally, twice daily) plus placebo Gefitinib (250 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: ASK120067; Drug: Placebo Gefitinib 250 mg
- Gefitinib + placebo ASK120067 (Active Comparator): Gefitinib (250 mg orally, once daily) plus placebo ASK120067 (80 mg orally, twice daily), in accordance with the randomization schedule.
  Interventions: Drug: Gefitinib; Drug: Placebo ASK120067

INTERVENTIONS:
Drug: ASK120067 — ASK120067 (80 mg orally twice daily) . A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: as long as patients are continuing to show clinical benefit according to RECIST 1.1, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: ASK120067+ placebo Gefitinib
Drug: Placebo Gefitinib 250 mg — The initial dose of Placebo Gefitinib 250 mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit according to RECIST 1.1, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Placebo Iressa 250 mg
  Arms: ASK120067+ placebo Gefitinib
Drug: Gefitinib — Gefitinib (250 mg orally, once daily) , A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: as long as patients are continuing to show clinical benefit acording to RECIST 1.1, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Gefitinib + placebo ASK120067
Drug: Placebo ASK120067 — Placebo ASK120067orally 80mg twice daily . A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit according to RECIST 1.1, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Gefitinib + placebo ASK120067

SUMMARY:
To assess the efficacy and safety of ASK120067 versus a standard of care epidermal growth factor receptor tyrosine kinase inhibitor Gefitinib in patients with locally advanced or Metastatic Non Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 18 years.
2. Histopathologically or pathologically confirmed adenocarcinoma of the lung.
3. Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy(including those with newly diagnosed or postoperative recurrent stage IIIb, IIIc, or IV cancer).
4. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R) that have been confirmed by the central laboratory testing report before enrollment (through tissue samples for testing cannot be derived from tumor lesions that have undergone radiotherapy, but can be obtained from newly developed lesions after local treatment) .
5. Patients must be treatment-naïve for locally advanced or metastatic NSCLC (excluding local treatment for non-target lesions) and eligible to receive first-line treatment. Prior adjuvant and neo-adjuvant therapy is permitted(chemotherapy, radiotherapy, investigational agents) if there is no disease progression one year after completion of treatment. Patients who have received local treatment (such as radiotherapy or pleural perfusion therapy) can participate in the study if the lesions covered by local treatment are non-target lesions.
6. At baseline, at least one tumor lesion must meet the following criteria:

   (i) It has not been previously treated with radiotherapy and has not been used for biopsy during the screening period; (ii) It can be accurately measured, with the longest diameter of ≥10 mm at baseline (lymph nodes must have a short axis of ≥15 mm); (iii) It can be assessed using both CT and MRI scans, but the same testing method must be used for subsequent evaluations.
7. Expected survival ≥ 3 months.
8. ECOG score of 0 to 1.
9. Reproductive-aged women must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result must be negative.
10. Reproductive-aged women should use strict contraceptive measures throughout the entire trial period and for 3 months after the last administration of the investigational drug. Male subjects should use strict contraceptive measures and should not engage in sperm donation throughout the entire trial period and for 6 months after the last administration of the investigational drug.
11. Provision of informed consent prior to any study specific procedures, sampling, and analysis.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior treatment with any systemic anti-cancer therapy for locally advanced/metastatic NSCLC;
   2. Prior treatment with an EGFR-TKI;
   3. Major surgery within 4 weeks of the first dose of study drug;
   4. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug;
   5. Patients currently (within 7 days before the first administration) receiving medications or herbal supplements known to be potent inducers of cytochrome P450 (CYP) 3A4;
   6. Neoadjuvant and adjuvant therapy (except in cases meeting the inclusion criterion 5);
   7. Patients who have received pleural infusion therapy must have stable pleural effusion for 28 days or more before they can be enrolled (intrapleural infusion therapy may use cytokines and immunostimulants, but not biological products or other drugs with long half-lives);
   8. Local radiotherapy or palliative radiotherapy for bone metastases within 14 days before the first administration of the investigational drug;
   9. Patients are receiving treatment with drugs that are known to prolong the QTc interval or potentially cause torsade de pointes, and require continued treatment with these drugs during the study;
   10. Discontinuation of other clinical trial drugs for less than 14 days prior to the first administration.
2. Patients with spinal cord compression or brain/meningeal metastases (except those who are asymptomatic, in stable condition, and do not require treatment with steroids for at least 4 weeks before the start of study treatment; patients who have received local radiotherapy for brain metastases must have remained stable for at least 28 days after radiotherapy before enrollment);
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
4. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of ASK120067.
5. Any of the following cardiac criteria:

   1. The average corrected (using the Fridericia formula) QT interval (QTcF), obtained from three resting electrocardiogram (ECG) examinations, is greater than 450 ms for males or 470 ms for females;
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG;
   3. Any patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval;
   4. Left ventricular ejection fraction (LVEF) ≤ 40%.
6. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
7. Patients with unrecovered toxic reactions of Grade 2 or above (based on the NCI-CTCAE 5.0 criteria) related to prior treatment at the start of the study treatment (excluding alopecia and Grade 2 neuropathy caused by platinum-based drugs).
8. Patients with mixed lung adenocarcinoma and squamous cell carcinoma.
9. Primary T790M+ patients.
10. Patients with poorly controlled hyperglycemia (when the fasting blood glucose is ≥7.0 mmol/L, the investigators should determine whether it can be stably controlled, and seek consultation with the endocrinology department if necessary).
11. Patients with inadequate bone marrow reserves or other organ dysfunctions, meeting any of the following criteria in laboratory tests (within 2 weeks before the laboratory blood drawing for the enrollment, no blood or blood products are transfused, and no granulocyte colony-stimulating factor or other hematopoietic stimulating factors are used for correction):

    1. Absolute neutrophil count<1.5×10^9/L;
    2. Platelet count <100 x 10^9/L;
    3. Hemoglobin <90 g/L;
    4. Alanine aminotransferase (ALT) or as aspartate aminotransferase (AST) levels >2.5 times the upper limit of normal in the absence of definitive hepatic metastases, or >5 times the upper limit of normal in the presence of hepatic metastases;
    5. Serum total bilirubin level > 1.5 times the upper limit of normal in the absence of definite hepatic metastases, or > 3 times the upper limit of normal in the presence of definite Gilbert syndrome (unconjugated hyperbilirubinemia) or hepatic metastases;
    6. Serum creatinine level >1.5 times.
12. Patients with a history of allergy or hypersensitivity to the active ingredient or inactive excipients of the investigational drug, drugs with chemical structures similar to the investigational drug, or drugs of the same class as the investigational drug.
13. Pregnant and lactating women.
14. Patients with other malignant tumors or diagnosed with other malignant tumors within the past 5 years (excluding clinically cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin, and papillary thyroid carcinoma).
15. Patients with any serious or uncontrolled ocular lesion that, in the judgment of the investigator, may bring an increased safety risk to them.
16. Subjects who, in the judgment of investigators, are not suitable for this study.
17. Involvement in the planning and/or conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  Progression-free survival was defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy prior to progression and was used to assess the efficacy of single agent ASK120067 compared with Gefitinib as measured by PFS.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  ORR was defined as the number (%) of patients with measurable disease with at least 1 visit response of Complete response (CR) or Partial response (PR) and it was used to further assess the efficacy of ASK120067 compared with Gefitinib defined as the number (%) of patients with measurable disease with at least 1 visit response of Complete response (CR) or Partial response (PR) and it was used to further assess the efficacy of ASK120067 compared with Gefitinib
Duration of Response (DoR) | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  Duration of response was defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression and was used to further assess the efficacy of ASK120067 compared with Gefitinib
Disease Control Rate (DCR) | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  The DCR was defined as the percentage of participants who had a best overall response (BOR) of Complete response (CR), Partial response (PR) or Stable disease (SD) ≥6 weeks prior to any Progressive disease (PD) event and was used to further assess the efficacy of ASK120067 compared with Gefitinib
Depth of Response | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  The Depth of response was defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions (TLs) at the nadir, in the absence of new lesions (NLs) or progression of Non-target lesions
Overall Survival (OS)- Number of Participants With an Event | Time from treatment start to the time of death due to any cause or withdrawal from study,whichever came first, assessed up to approximately 5 years
  Overall survival was defined as the time from the date of randomisation until death from any cause and was used to further assess the efficacy of ASK120067 compared with Gefitinib

OTHER OUTCOMES:
intracranial Progression-free survival (iPFS), intracranial Objective Response rate (iORR), intracranial duration of response (iDOR), intracranial Disease Control Rate (iDCR), and intracranial Depth of Response (iDepOR) | CT or MRI at screening and every 2 Cycles until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years
  For subjects with brain metastases at baseline, concurrent imaging examination of the brain lesion sites will be performed. Tumor response and PD will be additionally assessed by the Independent Review Committee (IRC) according to RECIST 1.1 criteria (for measurable lesions at baseline) for subjects with brain metastases at baseline.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

REFERENCES:
- [Derived] Shi Y, Wu L, Ji Y, Chen G, Li B, Bi M, Yang R, Miao L, Zhang G, Gao H, Sun L, Zhang M, Cang S, Sun M, Yao W, Pan Z, Cui J, Xiao Y, Wang Q; NCT04143607 Study Group. Efficacy and safety of limertinib versus gefitinib as first-line treatment for locally advanced or metastatic non-small-cell lung cancer with EGFR-sensitising mutation: a randomised, double-blind, double-dummy, phase 3 trial. Lancet Respir Med. 2025 Aug;13(8):677-686. doi: 10.1016/S2213-2600(25)00121-3. Epub 2025 Jun 20. PMID 40550238